CLINICAL TRIAL: NCT03742037
Title: A Phase 2b, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel Group Study to Evaluate the Efficacy, Safety, and Tolerability of Cenerimod in Subjects With Moderate to Severe Systemic Lupus Erythematosus (SLE)
Brief Title: Efficacy and Safety of Four Doses of Cenerimod Compared to Placebo in Adult Subjects With Active Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Viatris Innovation GmbH (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ID-064A202; 2018-001808-11 (EudraCT Number)
Record Dates: First submitted 2018-11-12; First posted 2018-11-15 (Actual); Results first posted 2023-09-22 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2023-09

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Musculoskeletal and connective tissue disorders
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Connective Tissue Diseases | interventions — cenerimod

STUDY DESIGN:
Intervention Model Description: Participants randomized to the 4 mg arm who are still on treatment at month 6 will be re-randomized in a 1:1 ratio to placebo or cenerimod 2 mg to enter Treatment Period 2 and will continue study treatment for a total maximum of 12 months.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Cenerimod 0.5 mg (Experimental): Participants will receive cenerimod 0.5 mg once daily in addition to background SLE therapy. Treatment Period 1 is 6 months long. It will start with the administration of the first dose of study treatment, after randomization, and end at the Month 6 visit. All randomized participants need to complete Treatment Period 1 before continuing in Treatment Period 2. In Treatment Period 2 participants will continue with cenerimod 0.5 mg for a further 6 months and end study treatment at the Month 12 visit.
  Interventions: Drug: Cenerimod 0.5 mg
- Cenerimod 1 mg (Experimental): Participants will receive cenerimod 1 mg once daily in addition to background SLE therapy. Treatment Period 1 is 6 months long. It will start with the administration of the first dose of study treatment, after randomization, and end at the Month 6 visit. All randomized participants need to complete Treatment Period 1 before continuing in Treatment Period 2. In Treatment Period 2 participants will continue with cenerimod 1 mg for a further 6 months and end study treatment at the Month 12 visit.
  Interventions: Drug: Cenerimod 1 mg
- Cenerimod 2 mg (Experimental): Participants will receive cenerimod 2 mg once daily in addition to background SLE therapy. Treatment Period 1 is 6 months long. It will start with the administration of the first dose of study treatment, after randomization, and end at the Month 6 visit. All randomized participants need to complete Treatment Period 1 before continuing in Treatment Period 2. In Treatment Period 2 participants will continue with cenerimod 2 mg for a further 6 months and end study treatment at the Month 12 visit.
  Interventions: Drug: Cenerimod 2 mg
- Cenerimod 2 mg (Ex-4mg) (Experimental): Half the participants that complete treatment with cenerimod 4 mg in Treatment Period 1 will be re-randomized to cenerimod 2 mg once daily in addition to background SLE therapy during Treatment Period 2. Participants will receive cenerimod 2 mg for 6 months and end study treatment at the Month 12 visit.
  Interventions: Drug: cenerimod 2 mg (ex-4 mg)
- Placebo (Ex-4mg) (Placebo Comparator): Half the participants that complete treatment with cenerimod 4 mg in Treatment Period 1 will be re-randomized to placebo (matching cenerimod) once daily in addition to background SLE therapy during Treatment Period 2. Participants will receive cenerimod 2 mg for 6 months and end study treatment at the Month 12 visit.
  Interventions: Drug: Placebo
- Cenerimod 4 mg (Experimental): Participants will received cenerimod 4 mg once daily in addition to background SLE therapy for up to 6 months in Treatment Period 1. The participants randomized to the 4 mg treatment who were still on treatment at Month 6 were re-randomized in a 1:1 ratio to placebo or cenerimod 2 mg to enter Treatment Period 2. The participants who did not complete 6 months of cenerimod 4 mg treatment will be analyzed in the "Non Re-randomized (Ex-4mg)" treatment group.
  Interventions: Drug: Cenerimod 4 mg
- Placebo (Placebo Comparator): Participants will receive placebo (matching cenerimod) once daily in addition to background SLE therapy. Treatment Period 1 is 6 months long. It will start with the administration of the first dose of study treatment, after randomization, and end at the Month 6 visit. All randomized participants need to complete Treatment Period 1 before continuing in Treatment Period 2. In Treatment Period 2 participants will continue with placebo (matching cenerimod) for a further 6 months and end study treatment at the Month 12 visit.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cenerimod 0.5 mg — Cenerimod will be supplied as a film-coated tablets at the dose of 0.5 mg
  Arms: Cenerimod 0.5 mg
Drug: Cenerimod 1 mg — Cenerimod will be supplied as a film-coated tablets at the dose of 1 mg
  Arms: Cenerimod 1 mg
Drug: Cenerimod 2 mg — Cenerimod will be supplied as a film-coated tablets at the dose of 2 mg
  Arms: Cenerimod 2 mg
Drug: Cenerimod 4 mg — Cenerimod will be supplied as a film-coated tablets at the dose of 4 mg
  Arms: Cenerimod 4 mg
Drug: Placebo — Matching placebo will be supplied as identical film-coated tablets formulated with the same excipients but without the active ingredient, cenerimod
  Arms: Placebo; Placebo (Ex-4mg)
Drug: cenerimod 2 mg (ex-4 mg) — Cenerimod will be supplied as a film-coated tablets at the dose of 2 mg
  Arms: Cenerimod 2 mg (Ex-4mg)

SUMMARY:
The purpose of the study is to assess the efficacy and safety of 4 doses of cenerimod versus placebo in adult subjects with systemic lupus erythematosus (SLE).

DETAILED DESCRIPTION:
This is a Phase 2b, multicenter, multinational, randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of 4 doses of cenerimod versus placebo in adult subjects with moderately to severely active, autoantibody-positive systemic lupus erythematosus (SLE).

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form prior to any study-mandated procedure
* Diagnosis of SLE made at least 6 months prior to Screening, by fulfilling at least 4 of the 11 criteria for SLE as defined by the American College of Rheumatology (ACR) criteria
* A mSLEDAI-2K score ≥ 6 of at least 2 points for musculoskeletal or mucocutaneous manifestations (i.e., myositis, arthritis, rash, alopecia, mucosal ulcers).
* Currently treated with stable doses of one or more of the following background medications:

  * NSAIDs
  * Anti-malarials (≤ 400 mg/day hydroxychloroquine, ≤ 500 mg/day chloroquine, ≤ 100 mg/day quinacrine)
  * Mycophenolate mofetil (≤ 2 g/day)
  * Mycophenolic acid (≤ 1440 mg/day)
  * Azathioprine (≤ 2 mg/kg/day)
  * Methotrexate (≤ 20 mg/week)
  * Corticosteroids (≤ 40 mg/day prednisone or equivalent)
  * Belimumab (≤10 mg/kg every 4 weeks intravenously, or 200 mg/week subcutaneously).
* History or presence of positive autoantibodies measured by central laboratory defined as follows: (a) Positive antinuclear antibody (ANA) test measured by immunofluorescence assay (IFA) with titre ≥1:80; AND/OR (b) positive anti-double stranded deoxyribonucleic acid (anti-dsDNA) antibodies with titre ≥30 IU/mL
* Women of childbearing potential:

  * Must have a negative serum pregnancy test at Screening
  * Must agree to undertake monthly urine pregnancy tests during the study
  * Must use highly effective methods of contraception from the screening visit until 6 months after taking the last dose of study treatment.

Exclusion Criteria:

* Active lupus nephritis or a renal biopsy demonstrating immune complex mediated glomerulonephritis compatible with lupus nephritis.
* CNS (Central Nervous System) lupus and severe forms of vasculitis requiring systemic immunosuppressive treatment
* A diagnosis of mixed connective tissue disease or any history of overlap syndromes of SLE with rheumatoid arthritis, erosive arthritis, scleroderma or autoimmune hepatitis
* History or presence of Mobitz type II or third-degree atrioventricular block, sick sinus syndrome, symptomatic bradycardia or syncope associated with cardiac disorders
* Subjects who experienced myocardial infarction, unstable angina pectoris, stroke, transient ischemic attack, vascular thrombosis, decompensated heart failure requiring hospitalization, or heart failure defined by the New York Heart Association Class III/IV within six months prior to Screening
* An elevated QT corrected for HR (Heart Rate) on the basis of Fridericia's formula interval of > 470 ms (females) / > 450 ms (males)
* History or presence of severe respiratory disease or pulmonary fibrosis
* Active or latent tuberculosis
* Ongoing bacterial, viral or fungal infection that is of clinical concern in the judgment of the investigator or history of any serious infection
* Subjects who have congenital or acquired severe immunodeficiency or known HIV infection or positive HIV testing
* Presence of macular edema or active uveitis
* Type 1 or 2 diabetes that is poorly controlled according to investigator judgment, or diabetes complicated with organ involvement such as diabetic nephropathy or retinopathy
* Significant hematology abnormality: Lymphocyte count < 800 /μL (0.8 × 10e9/L); hemoglobin < 9 g/dL; WBC (White Blood Cell) count < 2500/μL (2.5 × 10e9/L) or platelets < 75000/μL (75 × 10e9/L)
* Estimated glomerular filtration rate < 60 mL/min/1.73 m2
* Known allergy to S1P (sphingosine-1-phosphate) receptor modulators or any of the cenerimod formulation excipients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 427 (Actual)
Dates: Start 2018-12-21 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2022-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Viatris Innovation GmbH
Locations (148):
- United States (29):
  - Pinnacle Research Group, Anniston, Alabama
  - University of California San Diego, La Jolla, California
  - Valerius Medical Group and Research Center, Los Alamitos, California
  - University of Colorado School of Medicine, Aurora, Colorado
  - Robert W Levin MD PA, Clearwater, Florida
  - Center for Rheumatology Immunology and Arthritis, Fort Lauderdale, Florida
  - Life Clinical Trials, Margate, Florida
  - D&H National Research Centers INC, Miami, Florida
  - San Marcus Research Clinic, Miami Lakes, Florida
  - Millennium Research, Ormond Beach, Florida
  - Integral Rheumatology & Immunology Specialists, Plantation, Florida
  - Advanced Research Institute Inc Allergy & Rheumatology, St. Petersburg, Florida
  - Axiom Clinical Research of Florida, Tampa, Florida
  - North Georgia Rheumatology Group - Duluth, Lawrenceville, Georgia
  - Institute of Arthritis Research, Idaho Falls, Idaho
  - Washington University School of Medicine, St Louis, Missouri
  - Innovative Health Research, Las Vegas, Nevada
  - New York Presbyterian Columbia University Medical Center, New York, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Joint Muscle Medical Care and Research Institute - Lilington Office, Charlotte, North Carolina
  - DJL Clinical Research, Charlotte, North Carolina
  - Paramount Medical Research and Consulting, Middleburg Heights, Ohio
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Office of Ramesh C. Gupta, MD, Memphis, Tennessee
  - Amarillo Center for Clinical Research, Amarillo, Texas
  - Accurate Clinical Research, Houston, Texas
  - Southwest Rheumatology Research, LLC, Mesquite, Texas
  - Sun Research Institute, San Antonio, Texas
  - Accurate Clinical Management, Stafford, Texas
- Bulgaria (4):
  - Multiprofile Hospital For Active Treatment Trimontium, Plovdiv, Plodiv
  - University Multiprofile Hospital for Active Treatment Pulmed, Plovdiv
  - Diagnostic and Consulting Center "Aleksandrovska" EOOD, Sofia
  - Diagnostic Consulting Center Fokus-5, Sofia
- Chile (5):
  - Enroll SpA, Santiago
  - Biomedica Research Group, Santiago
  - Meditek Ltda., Santiago
  - Prosalud, Santiago
  - Clinical Research Chile SpA, Valdivia
- CCR Pardubice, Pardubice, Vychodocesky KRAJ, Czechia
- France (2):
  - Centre Hospitalier Regional Universitaire Brest Hôpital de la Cavale Blanche à Brest, Brest, Brittany Region
  - Hôpital Haut-Lévêque, Pessac
- Georgia (10):
  - LTD "New Plasma Clinic", Batumi
  - Aversi Clinic LTD, Tbilisi
  - Medi Club Georgia Ltd., Tbilisi
  - Ltd. Mtskheta Street Clinic, Tbilisi
  - The First Medical Center Ltd., Tbilisi
  - LLC "Innova", Tbilisi
  - LLC Raymann, Tbilisi
  - LTD "Tbilisi Heart Center", Tbilisi
  - Medicore, Tbilisi
  - Multiprofile Clinic Consilium Medulla, Tbilisi
- Städtisches Klinikum Karlsruhe gGmbH, Karlsruhe, Germany
- General Hospital of Athens "Laiko", Goudi, Greece
- Egyesitett Szent Istvan es Szent Laszlo Korhaz Rendelointezet, Budapest, Hungary
- Israel (4):
  - Rambam Healthcare Campus, Haifa
  - Bnai Zion Medical Center, Haifa
  - Galilee Medical Center, Nahariya
  - The Chaim Sheba Medical Center, Ramat Gan
- Italy (6):
  - LUPUS CLINIC c/o DIMI, Genova
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Ospedale San Raffaele, Milan
  - Azienda Ospedaliera San Camillo Forlanini, Roma
  - Fondazione Policlinico Universitario A. Gemelli, Roma
  - A.O. Mauriziano Umberto I di Torino, Torino
- Tomakomai City Hospital, Tomakomai-shi, Japan
- Mexico (18):
  - Consultorio Particular Dr. Miguel Cortés Hernández, Cuernavaca
  - Centro Integral en Reumatología S.A. de C.V., Guadalajara
  - Icle S.C., Guadalajara
  - Consultorio Privado de Especialidad del Dr. José Javier Orozco Alcalá, Guadalajara
  - Consultorio Médico del Dr. Federico Galván Villegas, Guadalajara
  - Morales Vargas Centro de Investigación S.C., León
  - Karla Adriana Espinosa Bautista, Mexico City
  - Centro de Investigación Clínica GRAMEL, S.C., Mexico City
  - Biológicos Especializados S.A. de C.V., Mexico City
  - Unidad de Atención Médica e Investigación en Salud, Mérida
  - Kohler & Milstein Research S.A. de C.V., Mérida
  - Accelerium, S. de R.L. de C.V., Monterrey
  - UBAM Unidad Biomédica Avanzada Monterrey, Monterrey
  - SMIQ, S. de R.L. de C.V., Querétaro
  - Hospital Universitario "Dr. Gonzalo Valdés Valdés", Saltillo
  - Unidad de Investigaciones Reumatológicas A.C., San Luis Potosí City
  - Centro de Atención e Investigación Cardiovascular del Potosí, S.C., San Luis Potosí City
  - Investigacion Biomedica para el Desarrollo de Farmacos S.A. de C.V., Zapopan
- Philippines (10):
  - Lipa Medix Medical Center, Lipa City, Batangas
  - Angeles University Foundation Medical Center, Angeles City
  - Davao Doctors Hospital, Davao City
  - Iloilo Doctors Hospital, Iloilo City
  - Makati Medical Center, Makati City
  - University of the Philippines Manila - Philippine General Hospital, Manila
  - Jose R. Reyes Memorial Medical Center, Manila
  - University of Santo Tomas Hospital, Manila
  - St. Luke's Medical Center, Quezon City
  - Far Eastern University - Nicanor Reyes Medical Foundation, Quezon City
- Poland (6):
  - Szpital Uniwersytecki Number 2 im. dr. Jana Biziela w Bydgoszczy, Bydgoszcz
  - Intermedius Uslugi Medyczne, Kościan
  - Szpital Specjalistyczny im. J. Dietla w Krakowie, Krakow
  - Centrum Medyczne Plejady, Krakow
  - Twoja Przychodnia Poznańskie Centrum Medyczne, Poznan
  - Śląskie Centrum Reumatologii, Rehabilitacji i Zapobiegania Niepełnosprawności im gen. Jerzego Zi, Ustroń
- Centro Reumatologico de Caguas, Caguas, Puerto Rico
- Romania (4):
  - Centrul Medical de Diagnostic si Tratament Ambulatoriu Neomed, Brasov
  - SC Sana Monitoring SRL, Bucharest
  - Spitalul Clinic "Sf. Maria", Bucharest
  - Spitalul Clinic Judetean de Urgenta Cluj-Napoca, Cluj-Napoca
- Russia (14):
  - Chelyabinsk Regional Clinical Hospital, Chelyabinsk
  - City Clinical Hospital #15 named after O.M. Filatova, Moscow
  - Federal State Budget Scientific Research Institution "Scientific Research Institute of Rheumatology n.a. V.A. Nasonova", Moscow
  - Non-governmental private healthcare organization, Scientific Clinical Centre of JSC Russian Railways, Moscow
  - Medical Center "Zdorovaya Semiya", LLC, Novosibirsk
  - Orenburg State Medical University, Orenburg
  - Clinical Rheumatological Hospital Number 25, Saint Petersburg
  - Military Medical Academy S.M. Kirov, Saint Petersburg
  - Polyclinic of Private Security and Detectives, Saint Petersburg
  - Medical Research Institute, LLC, Saint Petersburg
  - Medical Center Maksimum Zdorovia, Saint Petersburg
  - Saratov Regional Clinical Hospital, Saratov
  - State Institution of Health Protection "Clinical Hospital #8", Yaroslavl
  - JSC "Center of Family Medicine", Yekaterinburg
- Spain (5):
  - Hospital Universitario Regional de Málaga, Málaga, Malaga
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Quirónsalud Infanta Luisa, Seville
  - Hospital Universitario Doctor Peset, Valencia
- Taiwan (2):
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
- Thailand (2):
  - Rajavithi Hospital, Bangkok
  - Songklanagarind Hospital, Songkhla
- Turkey (Türkiye) (2):
  - Istanbul Universitesi Istanbul Tip Fakultesi, Istanbul
  - Necmettin Erbakan Üniversitesi Meram Tıp Fakültesi, Konya
- Ukraine (17):
  - Kyiv City Clinical Hospital №3, Kyiv
  - Clinic of State Institution "National Scientific Centre "Acad. Strazhesko Institute of Cardiology", Kyiv
  - Medical Centre "Consilium medical", Kyiv
  - Municipal Institution Kyiv Regional Council "Kyiv Regional Clinical Hospital", Kyiv
  - Municipal Nonprofit Institution of Lviv Regional Council "Lviv Regional Clinical Hospital", Lviv
  - Municipal Nonprofit Institution of Lviv Regional Council, Lviv
  - Lviv Regional Clinical Hospital, Lviv
  - Poltava Regional Clinical Hospital named after M.V. Sklifossovsky, Poltava
  - Ternopil University Clinic - Rheumatology department, Ternopil
  - Zakarpattya Regional Clinical Hospital n.a. A.Novak - Rheumatology Department, Uzhhorod
  - Private Small Scale Medical Center "Pulse", Vinnytsia
  - Medical Center "Health Clinic", LLC, Vinnytsia
  - Municipal Nonprofit Institution "Vinnytsia City Clinical Hospital №1", Vinnytsia
  - Vinnytsya Regional Clinical Hospital - Rheumatology Department, Vinnytsia
  - Scientific and Research Institute of Invalid Rehabilitation (EST Complex) of Vinnytsia M.I.Pyrogov NMU MOHU,, Vinnytsia
  - Municipal Institution "Zaporizhzhya Regional Clinical Hospital", Zaporizhzhya
  - Municipal institution "Regional Clinical Hospital n.a. O.F. Herbachevskoho", Zhytomyr
- United Kingdom (2):
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Guy's and Saint Thomas' NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Suffiotti M, Brazauskas P, Keller MP, Berkani O, Seifer G, Cornelisse P, Murphy MJ, Strasser DS. Pharmacodynamics of the S1P1 receptor modulator cenerimod in a phase 2b randomised clinical trial in patients with moderate to severe SLE. Ann Rheum Dis. 2025 Feb;84(2):284-293. doi: 10.1136/ard-2024-226547. Epub 2025 Jan 16. PMID 39919901
- [Derived] Askanase AD, D'Cruz D, Kalunian K, Merrill JT, Navarra SV, Cahuzac C, Cornelisse P, Murphy MJ, Strasser DS, Trokan L, Berkani O. Cenerimod, a sphingosine-1-phosphate receptor modulator, versus placebo in patients with moderate-to-severe systemic lupus erythematosus (CARE): an international, double-blind, randomised, placebo-controlled, phase 2 trial. Lancet Rheumatol. 2025 Jan;7(1):e21-e32. doi: 10.1016/S2665-9913(24)00246-7. Epub 2024 Nov 22. PMID 39586304

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was done from 21 December 2018 to 25 August 2022.
Pre-assignment Details: 427 participants are considered to be enrolled in the study and were randomized to study treatment. This represents the Full Analysis Set (treatment as assigned).
  810 adult subjects with SLE have been screened and 427 subjects randomized in a 1:1:1:1:1 ratio to placebo, 0.5, 1, 2, or 4 mg once daily (o.d.) of cenerimod, in addition to background SLE therapy.
Groups:
- Cenerimod 0.5 mg: Participants were randomized to receive cenerimod 0.5 mg once daily in addition to background SLE therapy for up to 6-months in Treatment Period 1. Participants completing Treatment Period 1 continued to receive cenerimod 0.5 mg once daily in addition to background SLE therapy during Treatment Period 2 for up to an additional 6 months. After end of treatment, participants entered a 6-month follow-up period.
- Cenerimod 1 mg: Participants were randomized to receive cenerimod 1 mg once daily in addition to background SLE therapy for up to 6-months in Treatment Period 1. Participants completing Treatment Period 1 continued to receive cenerimod 1 mg once daily in addition to background SLE therapy during Treatment Period 2 for up to an additional 6 months. After end of treatment, participants entered a 6-month follow-up period.
- Cenerimod 2 mg: Participants were randomized to receive cenerimod 2 mg once daily in addition to background SLE therapy for up to 6-months in Treatment Period 1. Participants completing Treatment Period 1 continued to receive cenerimod 2 mg once daily in addition to background SLE therapy during Treatment Period 2 for up to an additional 6 months. After end of treatment, participants entered a 6-month follow-up period.
- Cenerimod 2 mg (Ex-4 mg): Half the participants completing treatment with cenerimod 4 mg for up to 6-months in Treatment Period 1 were re-randomized to cenerimod 2 mg once daily in addition to background SLE therapy during Treatment Period 2. Participants received cenerimod 2 mg for up to 6 months. After end of treatment, participants entered a 6-month follow-up period.
- Placebo (Ex-4 mg): Half the participants completing treatment with cenerimod 4 mg for up to 6-months in Treatment Period 1 were re-randomized to placebo once daily in addition to background SLE therapy during Treatment Period 2. Participants received placebo for up to 6 months. After end of treatment, participants entered a 6-month follow-up period.
- Cenerimod 4 mg: Participants were randomized to receive cenerimod 4 mg once daily in addition to background SLE therapy for up to 6-months in Treatment Period 1. Participants randomized to the 4 mg treatment who were still on treatment at the end of Month 6 were re-randomized in a 1:1 ratio to placebo or cenerimod 2 mg to enter Treatment Period 2. After end of treatment, participants entered a 6-month follow-up period.
- Placebo: Participants were randomized to receive placebo once daily in addition to background SLE therapy for up to 6 months in Treatment Period 1. Participants completing Treatment Period 1 continued with placebo once daily in addition to background SLE therapy during Treatment Period 2 for up to an additional 6 months. After end of treatment, participants entered a 6-month follow-up period.
Period: Treatment Period 1 (1st Dose - Month 6)
Arm/Group | Cenerimod 0.5 mg | Cenerimod 1 mg | Cenerimod 2 mg | Cenerimod 2 mg (Ex-4 mg) | Placebo (Ex-4 mg) | Cenerimod 4 mg | Placebo
Started | 85 | 85 | 86 | 0 | 0 | 85 | 86
Completed | 78 | 78 | 71 | 0 | 0 | 70 | 77
Not Completed | 7 | 7 | 15 | 0 | 0 | 15 | 9
Not completed — Death | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 4 | 0 | 0 | 3 | 2
Not completed — Withdrawal by Subject | 4 | 1 | 2 | 0 | 0 | 2 | 4
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 1 | 0
Not completed — pre-specified criteria | 1 | 3 | 7 | 0 | 0 | 6 | 1
Not completed — Randomized but no study treatment taken | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Other reasons | 2 | 0 | 2 | 0 | 0 | 2 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 1
Period: Treatment Period 2 (Month 6 - Month 12)
Arm/Group | Cenerimod 0.5 mg | Cenerimod 1 mg | Cenerimod 2 mg | Cenerimod 2 mg (Ex-4 mg) | Placebo (Ex-4 mg) | Cenerimod 4 mg | Placebo
Started | 78 | 78 | 72 | 35 | 35 | 0 | 77
Completed | 74 | 74 | 59 | 30 | 35 | 0 | 68
Not Completed | 4 | 4 | 13 | 5 | 0 | 0 | 9
Not completed — Adverse Event | 1 | 2 | 3 | 1 | 0 | 0 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 2 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 2 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — pre-specified criteria | 0 | 1 | 3 | 2 | 0 | 0 | 2
Not completed — Other reasons | 2 | 0 | 2 | 0 | 0 | 0 | 1
Not completed — Discontinued study treatment in Treatment Period 1, re-randomized in error | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cenerimod 0.5 mg: Participants were randomized to receive cenerimod 0.5 mg once daily in addition to background SLE therapy for up to 6 months in Treatment Period 1.
- Cenerimod 1 mg: Participants were randomized to receive cenerimod 1 mg once daily in addition to background SLE therapy for up to 6 months in Treatment Period 1.
- Cenerimod 2 mg: Participants were randomized to receive cenerimod 2 mg once daily in addition to background SLE therapy for up to 6 months in Treatment Period 1.
- Cenerimod 4 mg: Participants were randomized to receive cenerimod 4 mg once daily in addition to background SLE therapy for up to 6 months in Treatment Period 1.
- Placebo: Participants were randomized to receive placebo once daily in addition to background SLE therapy for up to 6 months in Treatment Period 1.
- Total: Total of all reporting groups
Arm/Group | Cenerimod 0.5 mg | Cenerimod 1 mg | Cenerimod 2 mg | Cenerimod 4 mg | Placebo | Total
Number analyzed (Participants) | 85 | 85 | 86 | 85 | 86 | 427
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.8 (12.41) | 40.0 (12.77) | 42.2 (12.06) | 42.1 (10.44) | 41.0 (11.94) | 41.6 (11.94)
Age, Customized [Number; unit: years]
  Between 18 and 45 years | 49 | 54 | 49 | 50 | 57 | 259
  Between 45 and 64 years | 31 | 29 | 36 | 33 | 27 | 156
  Between 64 and 75 years | 5 | 2 | 1 | 2 | 2 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 83 | 80 | 82 | 82 | 406
  Male | 6 | 2 | 6 | 3 | 4 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 17 | 18 | 19 | 19 | 89
  Not Hispanic or Latino | 69 | 68 | 68 | 65 | 66 | 336
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 3 | 6 | 1 | 3 | 18
  Asian | 5 | 9 | 7 | 6 | 6 | 33
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 1
  Black or African American | 3 | 6 | 8 | 10 | 6 | 33
  White | 72 | 67 | 65 | 65 | 68 | 337
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  Bulgaria | 5 | 2 | 1 | 3 | 2 | 13
  Chile | 1 | 3 | 2 | 5 | 7 | 18
  Czechia | 2 | 2 | 2 | 0 | 1 | 7
  France | 0 | 0 | 0 | 1 | 0 | 1
  Georgia | 5 | 3 | 1 | 4 | 2 | 15
  Greece | 0 | 0 | 1 | 0 | 0 | 1
  Israel | 0 | 1 | 1 | 0 | 0 | 2
  Italy | 1 | 1 | 0 | 1 | 1 | 4
  Mexico | 10 | 6 | 10 | 6 | 7 | 39
  Philippines | 4 | 7 | 6 | 5 | 5 | 27
  Poland | 6 | 2 | 3 | 3 | 7 | 21
  Romania | 1 | 0 | 0 | 1 | 0 | 2
  Russia | 2 | 8 | 7 | 5 | 2 | 24
  Spain | 1 | 2 | 0 | 0 | 4 | 7
  Taiwan | 0 | 0 | 1 | 1 | 0 | 2
  Thailand | 0 | 2 | 0 | 0 | 0 | 2
  Turkey | 0 | 0 | 1 | 0 | 0 | 1
  Ukraine | 36 | 29 | 29 | 27 | 29 | 150
  United Kingdom | 0 | 0 | 0 | 2 | 1 | 3
  United States | 11 | 17 | 21 | 21 | 18 | 88
Body Mass Index [Mean (Standard Deviation); unit: kilograms/square meter] | 25.67 (5.67) | 25.55 (5.95) | 26.16 (6.6) | 26.82 (7.15) | 26.49 (6.24) | 26.14 (6.33)
modified SLEDAI at baseline [Mean (Standard Deviation); unit: units on a scale] — The SLEDAI-2K is a cumulative index of lupus disease activity. It is calculated from 24 individual descriptors across 9 organ systems, with weighted scores of 2-8. 0 points indicates inactive disease, and 105 points is the maximum possible score (Gladman D et al. J Rheumatol 2002;29;288-291). In this study the SLEDAI-2K was modified, to exclude leucopenia (minus 1 point), due to the mechanism of action of cenerimod. A score of 6 or greater is clinically relevant and associated with requiring lupus-directed therapy (Nuttall A et al. Best Pract Res Clin Rheumatol. 2013 Jun;27(3):309-18).
  units on a scale | 9.8 (2.69) | 10.1 (3.71) | 9.5 (2.88) | 10.0 (2.50) | 10.2 (3.05) | 9.9 (2.99)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Month 6 in the Modified Systemic Lupus Erythematosus Activity Index 2000 (mSLEDAI-2K) Score
Description: The primary endpoint is the absolute change from baseline in the modified Systemic Lupus Erythematosus Activity Index 2000 (mSLEDAI-2K) score. The SLEDAI-2K is a cumulative index of lupus disease activity scored by the physician. It is calculated from 24 individual descriptors across 9 organ systems, with weighted scores of 2-8, and measures disease activity within the last 10 days. 0 points indicates inactive disease, and 105 points is the maximum possible score. In this study the SLEDAI-2K was modified, to exclude leucopenia (minus 1 point), due to the mechanism of action of cenerimod. Improvement in systemic lupus erythematosus disease activity is defined as a reduction in SLEDAI-2K score of greater than or equal to 4. A decreased score, i.e., a negative change, indicates an improvement in systemic lupus erythematosus disease activity from baseline to Month 6.
Time Frame: Baseline (Day 1) and Month 6
Population: Full Analysis Set (FAS).
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Cenerimod 0.5 mg: Participants received cenerimod 0.5 mg once daily in addition to background SLE therapy for up to 6 months in treatment period 1.
- Cenerimod 1 mg: Participants received cenerimod 1 mg once daily in addition to background SLE therapy for up to 6 months in treatment period 1.
- Cenerimod 2 mg: Participants received cenerimod 2 mg once daily in addition to background SLE therapy for up to 6 months in Treatment Period 1.
- Cenerimod 4 mg: Participants received cenerimod 4 mg once daily in addition to background SLE therapy for up to 6-months in Treatment Period 1.
- Placebo: Participants received placebo, matching cenerimod, once daily in addition to SLE therapy for up to 6 months in Treatment Period 1.
Arm/Group | Cenerimod 0.5 mg | Cenerimod 1 mg | Cenerimod 2 mg | Cenerimod 4 mg | Placebo
Number analyzed (Participants) | 85 | 85 | 86 | 85 | 86
score on a scale | -3.2 [-3.98 to -2.49] | -3.41 [-4.16 to -2.67] | -2.84 [-3.58 to -2.09] | -4.04 [-4.79 to -3.28] | -2.85 [-3.60 to -2.10]
Statistical Analysis 1: Comparison: Cenerimod 0.5 mg vs Placebo; The analysis was performed on the Full Analysis Set (FAS). The FAS included all participants who were randomized. Baseline was defined as the last measurement before randomization; Test type: Superiority; p = 0.4749, Mixed Models Analysis; LS mean difference to placebo = -0.39, 95% CI 2-sided [-1.45 to 0.68], Standard Error of Mean 0.54
Statistical Analysis 2: Comparison: Cenerimod 1 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.2941, Mixed Models Analysis; LS mean to placebo = -0.57, 95% CI 2-sided [-1.65 to 0.49], Standard Error of Mean 0.54
Statistical Analysis 3: Comparison: Cenerimod 2 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.9802, Mixed Models Analysis; LS mean difference to placebo = 0.01, 95% CI 2-sided [-1.05 to 1.08], Standard Error of Mean 0.54
Statistical Analysis 4: Comparison: Cenerimod 4 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0291, Mixed Models Analysis; LS mean difference = -1.19, 95% CI 2-sided [-2.25 to -0.12], Standard Error of Mean 0.54

2. Secondary Outcome: Response on Systemic Lupus Erythematosus Responder Index 4 (SRI-4) at Month 6 as Compared to Baseline
Description: A responder could only be assessed if the full information of all body systems was available. A participant was defined as a responder based on the Systemic Lupus Erythematosus Responder Index 4 (SRI-4) was a composite, binary endpoint based on three variables:
  * mSLEDAI-2K score had to have a reduction from baseline greater than or equal to 4,
  * Physician Global Assessment (PGA) had to have an increase from baseline less than or equal to 0.3. The PGA is a 100 mm visual analog scale used by the physician to assess disease activity ranging for 0 to 3. The scale is anchored with values from 0 = "none" and 3 = "severe"), and
  * BILAG-2004 (no new BILAG A organ domain score and at most one new BILAG B organ domain score) compared with baseline.
  If one of the SRI-4 mSLEDAI-2K, PGA and BILAG variables were not met the subject was scored a non-responder. Participants that did not fit at least one of the above criteria were assigned to the missing group.
Time Frame: Baseline (Day 1) and Month 6
Population: Full Analysis Set (FAS)
Measure: Number; unit: participants
Groups:
- Cenerimod 4 mg: Participants received cenerimod 4 mg once daily in addition to background SLE therapy for up to 6 months in Treatment Period 1.
Arm/Group | Cenerimod 0.5 mg | Cenerimod 1 mg | Cenerimod 2 mg | Cenerimod 4 mg | Placebo
Number analyzed (Participants) | 85 | 85 | 86 | 85 | 86
participants
  Responder | 36 | 41 | 38 | 41 | 34
  Non-responder | 45 | 38 | 41 | 36 | 43
  Missing | 4 | 6 | 7 | 8 | 9
Statistical Analysis 1: Comparison: Cenerimod 0.5 mg vs Placebo; A generalized mixed effects model for repeated measures was applied to the SRI-4 response from Month 1 through 6 with treatment group, month, treatment group by month interaction, and stratification factors (oral corticosteroids dose & mSLEDAI-2K) as fixed effects & participant as random effect; Test type: Superiority; p = 0.974, Mixed Models Analysis; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.54 to 1.9]
Statistical Analysis 2: Comparison: Cenerimod 1 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.2845, Mixed Models Analysis; Odds Ratio (OR) = 1.42, 95% CI 2-sided [0.75 to 2.65]
Statistical Analysis 3: Comparison: Cenerimod 2 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.5115, Mixed Models Analysis; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.66 to 2.32]
Statistical Analysis 4: Comparison: Cenerimod 4 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.5115, Mixed Models Analysis; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.66 to 2.32]

3. Secondary Outcome: British Isles Lupus Assessment Group-2004 (BILAG) Disease Activity Index Response at Month 6
Description: The British Isles Lupus Assessment Group-2004 (BILAG) is a comprehensive tool used by the physician to assess disease activity and is sensitive to small changes over time.
  Response (no worsening) at Month 6 on BILAG-2004 disease activity index was defined as no new BILAG A organ domain score and no more than one new BILAG B organ domain score compared with baseline.
  No analysis is reported because the model did not meet the convergence criteria.
Time Frame: Baseline (Day 1) and Month 6
Population: Full analysis set (FAS).
Measure: Number; unit: percentage of participants
Arm/Group | Cenerimod 0.5 mg | Cenerimod 1 mg | Cenerimod 2 mg | Cenerimod 4 mg | Placebo
Number analyzed (Participants) | 81 | 79 | 79 | 77 | 77
percentage of participants | 98.8 | 98.7 | 97.5 | 98.7 | 97.4

ADVERSE EVENTS:
Time Frame: Treatment-emergent Adverse Events (TEAEs) are reported. TEAEs are defined as adverse events with onset on or after the date of first intake of double-blind study treatment up to end of treatment plus 6 months (i.e., maximum of 18 months: Treatment Period 1 + Treatment Period 2 + 6-month safety follow-up period). Subjects who received cenerimod 4 mg and completed Treatment Period 1 were re-randomized to cenerimod 2 mg or placebo in Treatment Period 2.
Description: TEAEs are reported for the Safety Analysis Set, i.e., according to the actual treatment received, which may have differed from the assigned study treatment (see Participant Flow, above). Note that 1 subject was randomized to the cenerimod 0.5 mg arm/group but received cenerimod 2 mg during Treatment Period 2. This subject is thus included in the 'at risk' population of the cenerimod 2 mg arm/group (n = 87) and not in the cenerimod 0.5 mg arm/group (n = 84) for the reporting of TEAEs.
Groups:
- Cenerimod 0.5 mg (Treatment Period 1 & 2): Participants received cenerimod 0.5 mg once daily in addition to background SLE therapy for up to 6 months in Treatment Period 1. Participants completing Treatment Period 1 continued with cenerimod 0.5 mg once daily in addition to background SLE therapy during treatment period 2 for up to an additional 6 months. After end of treatment, participants entered a 6-month follow-up period.
- Cenerimod 1 mg (Treatment Period 1 & 2): Participants received cenerimod 1 mg once daily in addition to background SLE therapy for up to 6 months in Treatment Period 1. Participants completing Treatment Period 1 continued to receive cenerimod 1 mg once daily in addition to background SLE therapy during Treatment Period 2 for up to an additional 6 months. After end of treatment, participants entered a 6-month follow-up period.
- Cenerimod 2 mg (Treatment Period 1 & 2): Participants received cenerimod 2 mg once daily in addition to background SLE therapy for up to 6 months in treatment period 1. Participants completing Treatment Period 1 continued to receive cenerimod 2 mg once daily in addition to background SLE therapy during Treatment Period 2 for up to an additional 6 months. After end of treatment, participants entered a 6-month follow-up period.
- Cenerimod 4 mg (Treatment Period 1) & Cenerimod 2 mg (Ex-4 mg; Treatment Period 2): Half the participants completing treatment with cenerimod 4 mg in Treatment Period 1 were re-randomized to cenerimod 2 mg once daily in addition to background SLE therapy during Treatment Period 2. Participants received cenerimod 2 mg for up to 6 months. After end of treatment, participants entered a 6-month follow-up period.
- Cenerimod 4 mg (Treatment Period 1) & Placebo (Ex-4 mg; Treatment Period 2): Half the participants completing treatment with cenerimod 4 mg in Treatment Period 1 were re-randomized to placebo once daily in addition to background SLE therapy during Treatment Period 2. Participants received placebo for up to 6 months. After end of treatment, participants entered a 6-month follow-up period.
- Cenerimod 4 mg (Treatment Period 1) & Not Re-randomized (Ex-4 mg; Treatment Period 2): Participants were not re-randomized and did not receive treatment in Treatment Period 2. (These participants previously received cenerimod 4 mg once daily in addition to background SLE therapy for 6 months in treatment period 1). After end of treatment, participants entered a 6-month follow-up period.
- Placebo (Treatment Period 1 & 2): Participants received placebo once daily in addition to background SLE therapy for up to 6 months in Treatment Period 1. Participants completing Treatment Period 1 continued with placebo once daily in addition to background SLE therapy during Treatment Period 2 for up to an additional 6 months. After end of treatment, participants entered a 6-month follow-up period.
Arm/Group | Cenerimod 0.5 mg (Treatment Period 1 & 2) | Cenerimod 1 mg (Treatment Period 1 & 2) | Cenerimod 2 mg (Treatment Period 1 & 2) | Cenerimod 4 mg (Treatment Period 1) & Cenerimod 2 mg (Ex-4 mg; Treatment Period 2) | Cenerimod 4 mg (Treatment Period 1) & Placebo (Ex-4 mg; Treatment Period 2) | Cenerimod 4 mg (Treatment Period 1) & Not Re-randomized (Ex-4 mg; Treatment Period 2) | Placebo (Treatment Period 1 & 2)
All-Cause Mortality (participants affected / at risk) | 0/84 | 2/85 | 0/87 | 0/35 | 0/35 | 0/14 | 0/86
Serious Adverse Events (participants affected / at risk) | 4/84 | 12/85 | 4/87 | 1/35 | 0/35 | 2/14 | 6/86
Other Adverse Events (participants affected / at risk) | 37/84 | 54/85 | 53/87 | 23/35 | 20/35 | 13/14 | 39/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cenerimod 0.5 mg (Treatment Period 1 & 2) (N=84) | Cenerimod 1 mg (Treatment Period 1 & 2) (N=85) | Cenerimod 2 mg (Treatment Period 1 & 2) (N=87) | Cenerimod 4 mg (Treatment Period 1) & Cenerimod 2 mg (Ex-4 mg; Treatment Period 2) (N=35) | Cenerimod 4 mg (Treatment Period 1) & Placebo (Ex-4 mg; Treatment Period 2) (N=35) | Cenerimod 4 mg (Treatment Period 1) & Not Re-randomized (Ex-4 mg; Treatment Period 2) (N=14) | Placebo (Treatment Period 1 & 2) (N=86)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic mass (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral toxoplasmosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Systemic lupus erythematosus rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertensive emergency (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cenerimod 0.5 mg (Treatment Period 1 & 2) (N=84) | Cenerimod 1 mg (Treatment Period 1 & 2) (N=85) | Cenerimod 2 mg (Treatment Period 1 & 2) (N=87) | Cenerimod 4 mg (Treatment Period 1) & Cenerimod 2 mg (Ex-4 mg; Treatment Period 2) (N=35) | Cenerimod 4 mg (Treatment Period 1) & Placebo (Ex-4 mg; Treatment Period 2) (N=35) | Cenerimod 4 mg (Treatment Period 1) & Not Re-randomized (Ex-4 mg; Treatment Period 2) (N=14) | Placebo (Treatment Period 1 & 2) (N=86)
Lymphopenia (Blood and lymphatic system disorders) | 4 (4) | 10 (12) | 12 (18) | 7 (12) | 4 (4) | 5 (7) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 4 (7) | 1 (1) | 1 (1) | 2 (4) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Cataract subcapsular (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 3 (3) | 2 (2) | 9 (9) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Eye irritation (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 6 (6) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Acid peptic disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (6) | 4 (6) | 3 (4) | 3 (4) | 0 (0) | 0 (0) | 3 (4)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (3) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 8 (8) | 8 (9) | 10 (10) | 1 (1) | 2 (2) | 2 (2) | 11 (11)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Eyelid infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 5 (5) | 0 (0) | 6 (6) | 3 (3) | 1 (1) | 1 (1) | 5 (5)
Ophthalmic herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 2 (5) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 2 (2) | 2 (5) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (2)
Upper respiratory tract infection (Infections and infestations) | 7 (8) | 4 (5) | 5 (5) | 4 (4) | 2 (2) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 2 (2) | 2 (2) | 4 (4) | 0 (0) | 1 (1) | 9 (9)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bone contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 5 (7) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Forced expiratory volume decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Liver function test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 1 (2) | 2 (2) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 4 (6) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Osteitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 4 (8)
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 11 (12) | 12 (13) | 8 (9) | 8 (10) | 2 (2) | 1 (1) | 4 (5)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Brachioradial pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Macule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 8 (8) | 3 (3) | 8 (10) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any study-related publication written independently by investigators must be submitted to the sponsor for review at least 30 days prior to submission for publication or presentation.

Upon review, the sponsor may provide comments and may also request alterations and/or deletions for the sole purpose of protecting its confidential information and/or patent rights. Neither the institution nor the investigator should permit publication during such a review period.

DOCUMENTS (3):
  • Study Protocol: Protocol (2022-02-04): https://cdn.clinicaltrials.gov/large-docs/37/NCT03742037/Prot_000.pdf
  • Study Protocol: COVID-19 addendum to protocol (2020-05-27): https://cdn.clinicaltrials.gov/large-docs/37/NCT03742037/Prot_001.pdf
  • Statistical Analysis Plan (2022-09-27): https://cdn.clinicaltrials.gov/large-docs/37/NCT03742037/SAP_002.pdf